CLINICAL TRIAL: NCT04012775
Title: An Open-label, Randomized, Multi-center, Parallel-group Clinical Trial Comparing the Efficacy and Safety of Rinsulin® NPH ("Geropharm", Russia) With Humulin® NPH ("Lilly France", France) in Type 2 Diabetes Mellitus Patients
Brief Title: Efficacy and Safety of Insulin Rinsulin® NPH Compared to Humulin® NPH in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RINPH-IM
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin Humulin® NPH (Active Comparator): Insulin Humulin® NPH twice daily, individually glucose-level based administered doses +/- 1,2 or 3 OADs in stable doses, started before enrollment
  Interventions: Biological: Insulin Humulin® NPH
- Insulin Rinsulin® NPH (Experimental): Insulin Rinsulin® NPH twice daily, individually glucose-level based administered doses +/- 1,2 or 3 OADs in stable doses, started before enrollment
  Interventions: Biological: Insulin Rinsulin® NPH

INTERVENTIONS:
Biological: Insulin Humulin® NPH — 4 weeks of glucose-level based dose titration, 24 weeks of treatment with stable doses
  Arms: Insulin Humulin® NPH
Biological: Insulin Rinsulin® NPH — 4 weeks of glucose-level based dose titration, 24 weeks of treatment with stable doses
  Arms: Insulin Rinsulin® NPH

SUMMARY:
The study is designed to approve non-inferior efficacy and safety of Rinsulin® NPH compared to Humulin® NPH.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent
* Diabetes mellitus type 2
* Indications for Rinsulin NPH / Humalog NPH treatment
* Glycosylated hemoglobin (HbA1c) level of 6.5 to 12.0 % at screening (both values inclusive)
* Body mass index (BMI) of 18.0 to 35 kg/m2 at screening (both values inclusive).
* Female patients of childbearing potential who are willing to use two acceptable methods of contraception, (e.g., intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.), from the time of screening and for the duration of the trial, through trial completion.

Exclusion Criteria:

* Age less than 18 years old at screening
* Pregnant and breast-feeding women
* Need of administration of glucocorticoid therapy or any other therapy that may influence glucose level
* Administration of any immunosupressive drugs (Cyclosporinum, Methotrexatum)
* Serological evidence of human immunodeficiency virus (HIV), hepatitis B (HbSAg), hepatitis C (HCVAb) or antibodies to Treponema pallidum (syphilis) at screening.
* History of hypersensitivity to any of the active or inactive ingredients of the insulin/insulin analogue preparations used in the trial, OR history of significant allergic drug reactions.
* History of hematological disorders that can affect the reliability of HbA1c estimation (hemoglobinopathies, hemolytic anemia, etc.).
* History or presence of a medical condition or disease that in the investigator's opinion would embarrass glycemic control and completion of the study
* Presence of severe diabetes complications
* Receipt of another investigational drug in the 3 months prior to screening
* Acute psychiatric disorder or exacerbation of chronic psychiatric disorder at screening
* History or presence of drug abuse
* Positive test for addictive substance in urine at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
Antibody Response | 24 weeks
  Change from baseline in titer of antibodies to human insulin

SECONDARY OUTCOMES:
Hypoglycemic episodes (glucose level < 3.9 mmol/l) frequency | 28 weeks (4 + 24 weeks)
Change in BMI from baseline | 24 weeks
Occurrence of adverse events | 28 weeks (4 + 24 weeks)
Occurrence of Injection Site Reaction | 28 weeks (4 + 24 weeks)
Change in HbA1c from baseline | 24 weeks
Change in fasting plasma glucose level from baseline | 4 weeks
Change in fasting plasma glucose level from baseline | 16 weeks
Change in fasting plasma glucose level from baseline | 28 weeks
Change in basal insulin dose per body weight (U/kg) from baseline | 24 weeks
Change in total basal insulin dose (U) from baseline | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Olga A Miroshnichenko, PhD, Principal Investigator — Saint Petersburg State Diagnostic Center № 85
Locations (14):
- Russia (14):
  - Chelyabinsk Railway Clinical Hospital, Chelyabinsk
  - Moscow Endocrinological Dispensary, Moscow
  - Moscow Clinical Hospital № 71, Moscow
  - Nizhny Novgorod Regional Clinical Hospital, Nizhny Novgorod
  - V.A. Baranov Republic Hospital, Petrozavodsk
  - City Polyclinic № 6, Saint Petersburg
  - City Hospital № 2, Saint Petersburg
  - City Polyclinic № 17, Saint Petersburg
  - Medical Sanitary Unit № 157, Saint Petersburg
  - Institute of Medical Research, Saint Petersburg
  - Research Center Eco-Safety, Saint Petersburg
  - Saint Petersburg State Diagnostic Center № 85, Saint Petersburg
  - Diabetes Center, Samara
  - Clinical Hospital № 3, Yaroslavl

IPD SHARING:
Plan to Share IPD: No